CLINICAL TRIAL: NCT01227785
Title: Next Generation INCEPTA ICD and CRT-D Field Following Study: Respiratory Rate Trend Evaluation in Heart Failure (HF) Patients
Brief Title: Next Generation INCEPTA Implantable Cardioverter Defibrillator (ICD) and Cardiac Resynchronization Therapy (CRT-D) Field Following Study
Acronym: NOTICE-HF
Status: Completed | Type: Observational
Sponsor: Guidant Corporation (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: NOTICE-HF 0410
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Sudden Cardiac Death; Heart Failure
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- INCEPTA ICD and CRT-D: ICD and CRT-D indicated patients were included in the study. Overall patient population, CRT-D or ICD populations, and patients experiencing or not experiencing a protocol-defined heart failure event were included (dependent on outcomes measured).
  Interventions: Device: INCEPTA ICD or CRT-D

INTERVENTIONS:
Device: INCEPTA ICD or CRT-D

SUMMARY:
This study has 2 purposes:

The first purpose of the study is to test a new family of Boston Scientific Implantable Cardioverter Defibrillators ("ICDs") and cardiac resynchronization therapy ICDs ("CRT-Ds") and show how well these new devices work in patients. This new family is called the INCEPTA ICD and the INCEPTA CRT-D.

The second purpose of the study is to collect data from a feature that monitors breathing. It is called the Respiratory Rate Trend (RRT). These data will help to better understand how changes in breathing relate to changes in clinical conditions.

DETAILED DESCRIPTION:
Study Purpose

Study purpose I:

To evaluate and document appropriate clinical performance of the INCEPTA (DR and VR) implantable cardioverter defibrillator (ICD) system and the INCEPTA cardiac resynchronization therapy ICD (CRT-D) system and associated application software.

Study purpose II:

Demonstrate the clinical relevance of chronic ambulatory daily median Respiratory Rate Trend (RRT) in HF patients

Study Device

* INCEPTA (DR and VR) implantable cardioverter defibrillator (ICD) system (Models F160, F161, F162, F163)
* INCEPTA cardiac resynchronization therapy ICD (CRT-D) system (Models P162, P163, P165)

Indication ICD / CRT-D Indication according to standard clinical practice

Study Objectives

The study has two primary objectives, linked to the respective study purposes:

For purpose I:

The objective is to collect data on the clinical performance of the INCEPTA ICD and CRT-D devices during standard clinical use at implant, pre-discharge and at a 1-month post-implant. Clinical performance included analysis of pacing thresholds, pacing impedance, sensing thresholds, number of successfully converted VT/VF episodes, induced episodes detection times, spontaneous episodes, wanded telemetry, adverse events (AEs) and product experiences.

For purpose II:

The objective is to show that daily median respiratory rate increases more in patients who experience an HF-event (Group 1) than in patients who do not experience an HF-event (Group 2).

This is a prospective, multi-centre, field following study.

Up to 35 study centers in the International geography will enrol 120 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing and capable of providing informed consent, undergoing a device implant, participating in all testing associated with this clinical study;
* Patients whose age is 18 or above, or of legal age to give informed consent specific to national law
* Patients indicated for an ICD according to normal clinical practice (for those patients receiving an INCEPTA ICD).

  -As soon as 20 ICD patients are included in the study for purpose I, only NYHA Class III patients will be allowed in the study.
* New York Heart Association (NYHA) Class III patients indicated for a CRT-D according to normal clinical practice (for those patients receiving an INCEPTA CRT-D).

Exclusion Criteria:

* Women of childbearing potential who are or might be pregnant at the time of the study (method of assessment upon physician's discretion)
* Enrolled in any other concurrent study.
* Inability or refusal to comply with the follow-up schedule
* Patients that have received routinely scheduled intravenous inotropic therapy as part of their drug regimen within the past 90 days
* Patients prescribed to positive airway pressure therapy
* A life expectancy of less than 1 year, per physician discretion
* Patient in NYHA Class IV during the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients should be selected from the investigator's general population and be indicated for an ICD or CRT-D implantation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum Berlin, Berlin, State of Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: Nov2010 - Feb2011
Groups:
- INCEPTA ICD and CRT-D: Patients implanted with Incepta ICD or CRT-D device
Period: Overall Study
Arm/Group | INCEPTA ICD and CRT-D
Started | 120
Completed | 108
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | INCEPTA ICD and CRT-D
Number analyzed (Participants) | 120
Age, Customized [Mean (Standard Deviation); unit: years]
  ICD | 62.7 (10.6)
  CRT-D | 67.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 100

OUTCOME MEASURES:

1. Primary Outcome: Clinical Performance for Left Ventricular (LV) Sensing Amplitude at Implant for CRT-D Patients
Description: Left Ventricular (LV) Sensed Amplitude results were reported at implant for CRT-D patients.
Time Frame: implant
Population: The number of CRT-D patients with available data at implant
Measure: Mean (Standard Deviation); unit: milli volt (mV)
Arm/Group | INCEPTA CRT-D Patients
Number analyzed (Participants) | 74
milli volt (mV) | 14.4 (7.3)

2. Secondary Outcome: Evaluate the Daily Median Respiratory Rate Trend in Patients Who Experience a HF-event Compared to Patients Who do Not Experience a HF-event.
Description: A comparison of the change in respiratory rate trend over time was made between patients who experienced a protocol-defined HF event (HFE) (Group1: Patients with a HFE) and patients who did not experience a protocol-defined heart failure event (Group 2: Patients without a HFE). Only patients with at least 3 valid daily respiratory rate values (60%) out of each 5-day window were evaluated. The objective was to show that daily median respiratory rate increases more in patients who experience a HFE (Group 1) than in patients who do not experience an HFE (Group 2). A comparison between patients who experience a HFE (Group 1) and patients who do not experience a HFE (Group 2). Two average daily median respiratory rates were done per patient: 60 to 56 days before an index time and 11 to 7 days before the same index time; the difference between these two averaged daily median respiratory rates was done. Index time=day of the first HFE (Group 1) and day of 6-month visit (Group 2).
Time Frame: Results were captured from implant time window to the first event for patients with HFE, up to an average of 9 months
Population: HF events were reported and adjudicated to classify patients into group 1 or 2. Group 1=17 HFEs in 13 patients. For patients with multiple HFEs,only the first with sufficient data was used. 8/13 with a HFE had data for the endpoint analysis.Group 2=95 patients with 9 month follow-up. 90/95 had data eligible for inclusion in the endpoint analysis.
Measure: Median (Inter-Quartile Range); unit: breaths/min
Groups:
- Group1: Patients With a HFE: Patients who experienced a protocol-defined HF event
- Group 2: Patients Without a HFE: Patients who did not experience a protocol-defined HFE
Arm/Group | Group1: Patients With a HFE | Group 2: Patients Without a HFE
Number analyzed (Participants) | 8 | 90
breaths/min | -0.30 [-0.47 to 0.30] | 0 (1.06) [-0.40 to 0.80]

3. Primary Outcome: Clinical Performance at Pre-discharge for LV Sensing Amplitude for CRT-D Patients
Description: Left Ventricular (LV) Sensed Amplitude results were reported pre-discharge for CRT-D patients.
Time Frame: pre-discharge
Population: 69 patients in the CRT-D arm had available data at pre-discharge visit.
Measure: Mean (Standard Deviation); unit: milli volt (mV)
Arm/Group | INCEPTA CRT-D Patients
Number analyzed (Participants) | 69
milli volt (mV) | 14.9 (7.7)

4. Primary Outcome: Clinical Performance at1-month for Left Ventricular (LV) Sensing Amplitude for CRT-D Patients
Description: LV Sensed Amplitude results were reported at 1-month post-implant for CRT-D patients.
Time Frame: 1-month
Population: 68 patients in the CRT-D cohort had available data at 1month visit
Measure: Mean (Standard Deviation); unit: milli volt (mV)
Arm/Group | INCEPTA CRT-D Patients
Number analyzed (Participants) | 68
milli volt (mV) | 17.2 (7.1)

5. Primary Outcome: Clinical Performance at Implant for Right Atrium (RA) Sensing Amplitude
Description: RA Sensed Amplitude results were reported for implant for CRT-D and ICD patients
Time Frame: implant
Population: 55 CRT-D patients and 11 ICD patients had available data at implant.
Measure: Mean (Standard Deviation); unit: milli volt (mV)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 55 | 11
milli volt (mV) | 3.8 (2.0) | 3.2 (2.2)

6. Primary Outcome: Clinical Performance at Pre-discharge for RA Sensing Amplitude
Description: RA Sensed Amplitude results were reported at pre-discharge for CRT-D and ICD patients
Time Frame: pre-discharge
Population: 55 CRT-D and 11 ICD patients had data available at pre-discharge visit.
Measure: Mean (Standard Deviation); unit: milli volt (mV)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 55 | 11
milli volt (mV) | 4.1 (2.0) | 3.9 (2.6)

7. Primary Outcome: Clinical Performance at1-month for RA Sensing Amplitude
Description: RA Sensed Amplitude results were reported at 1-month post-implant for CRT-D and ICD patients
Time Frame: 1-month
Population: 53 CRT-D and 11 ICD patients had data available at 1-month visit.
Measure: Mean (Standard Deviation); unit: milli volt (mV)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 53 | 11
milli volt (mV) | 4.9 (2.9) | 3.7 (2.7)

8. Primary Outcome: Clinical Performance at Implant for Right Ventricle (RV) Sensing Amplitude
Description: RV Sensed Amplitude results were reported at implant for CRT-D and ICD patients
Time Frame: implant
Population: 74 CRT-D and 45 ICD patients had data available at implant
Measure: Mean (Standard Deviation); unit: milli volt (mV)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 74 | 45
milli volt (mV) | 16.2 (6.6) | 15.8 (5.8)

9. Primary Outcome: Clinical Performance at Pre-discharge for Right Ventricle (RV) Sensing Amplitude
Description: RV Sensed Amplitude results were reported at pre-discharge for CRT-D and ICD patients
Time Frame: pre-discharge
Population: 73 CRT-D and 44 ICD patients had data available at pre-discharge visit.
Measure: Mean (Standard Deviation); unit: milli volt (mV)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 73 | 44
milli volt (mV) | 16.7 (6.1) | 16.9 (5.9)

10. Primary Outcome: Clinical Performance at1-month for Right Ventricle (RV) Sensing Amplitude
Description: RV Sensed Amplitude results were reported at 1-month post-implant for CRT-D and ICD patients
Time Frame: 1month
Population: 68 CRT-D and 43 ICD patients had data available at 1month visit.
Measure: Mean (Standard Deviation); unit: milli volt (mV)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 68 | 43
milli volt (mV) | 17.9 (6.2) | 17.1 (16.6)

11. Primary Outcome: Clinical Performance at Implant for LV Pacing Threshold
Description: LV pacing threshold results were reported for CRT-D patients at implant.
Time Frame: implant
Population: 78 CRT-D patients had data available at implant.
Measure: Mean (Standard Deviation); unit: volts (V)
Arm/Group | INCEPTA CRT-D Patients
Number analyzed (Participants) | 78
volts (V) | 1.3 (0.8)

12. Primary Outcome: Clinical Performance at Pre-discharge for LV Pacing Threshold
Description: LV pacing threshold results were reported at pre-discharge for CRT-D patients.
Time Frame: pre-discharge
Population: 75 patients had data available at pre-discharge
Measure: Mean (Standard Deviation); unit: volts (V)
Arm/Group | INCEPTA CRT-D Patients
Number analyzed (Participants) | 75
volts (V) | 1.5 (1.2)

13. Primary Outcome: Clinical Performance at1-month for LV Pacing Threshold
Description: LV pacing threshold results were reported at 1-month post-implant for CRT-D patients.
Time Frame: 1-month
Population: 73 CRT-D patients had data available at 1-month visit.
Measure: Mean (Standard Deviation); unit: volts (V)
Arm/Group | INCEPTA CRT-D Patients
Number analyzed (Participants) | 73
volts (V) | 1.3 (0.9)

14. Primary Outcome: Clinical Performance at Implant for RV Pacing Threshold
Description: RV pacing threshold results were reported at implant
Time Frame: implant
Population: 79 CRT-D and 46 ICD patients had data available at implant.
Measure: Mean (Standard Deviation); unit: volts (V)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 79 | 46
volts (V) | 0.7 (0.3) | 0.8 (0.5)

15. Primary Outcome: Clinical Performance at Pre-discharge for RV Pacing Threshold
Description: RV pacing threshold results were reported at pre-discharge
Time Frame: pre-discharge
Population: 78 CRT-D and 45 ICD patients had data available at pre-discharge
Measure: Mean (Standard Deviation); unit: volts (V)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 78 | 45
volts (V) | 0.7 (0.3) | 0.8 (1.1)

16. Primary Outcome: Clinical Performance at 1-month for RV Pacing Threshold
Description: RV pacing threshold results were reported at 1-month post-implant
Time Frame: 1-month
Population: 75 CRT-D and 43 ICD patients had data available at 1-month visit.
Measure: Mean (Standard Deviation); unit: volts (V)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 75 | 43
volts (V) | 0.9 (0.5) | 1.4 (1.7)

17. Primary Outcome: Clinical Performance at Implant for RA Pacing Threshold
Description: RA pacing threshold results were reported for implant
Time Frame: implant
Population: 56 CRT-D and 11 ICD patients had data available at implant
Measure: Mean (Standard Deviation); unit: volts (V)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 56 | 11
volts (V) | 0.8 (0.7) | 1.0 (0.7)

18. Primary Outcome: Clinical Performance at Pre-discharge for RA Pacing Threshold
Description: RA pacing threshold results were reported at pre-discharge
Time Frame: pre-discharge
Population: 57 CRT-D and 11 ICD patients had data available at pre-discharge
Measure: Mean (Standard Deviation); unit: volts (V)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 57 | 11
volts (V) | 0.8 (0.9) | 0.9 (0.8)

19. Primary Outcome: Clinical Performance at 1-month for RA Pacing Threshold
Description: RA pacing threshold results were reported at 1-month post-implant
Time Frame: 1-month
Population: 54 CRT-D and 11 ICD patients had data available at 1-month visit
Measure: Mean (Standard Deviation); unit: volts (V)
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 54 | 11
volts (V) | 1.0 (1.0) | 1.0 (0.7)

20. Primary Outcome: Clinical Performance at Implant LV Pacing Impedance for CRT-D.
Description: LV pacing impedance results at implant were measured in CRT-D.
Time Frame: implant
Population: 78 CRT-D patients had data available at implant
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | INCEPTA CRT-D Patients
Number analyzed (Participants) | 78
Ohms | 879 (296)

21. Primary Outcome: Clinical Performance at Pre-discharge for LV Pacing Impedance for CRT-D.
Description: LV pacing impedance results were reported for pre-discharge visit
Time Frame: pre-discharge
Population: 75 CRT-D patients had data available at pre-discharge
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | INCEPTA CRT-D Patients
Number analyzed (Participants) | 75
Ohms | 777 (244)

22. Primary Outcome: Clinical Performance at 1-month for LV Pacing Impedance for CRT-D.
Description: LV pacing impedance results were reported at 1-month post-implant
Time Frame: 1-month
Population: 73 CRT-D patients had data available at 1-month visit
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | INCEPTA CRT-D Patients
Number analyzed (Participants) | 73
Ohms | 778 (265)

23. Primary Outcome: Clinical Performance at Implant for RV Pacing Impedance
Description: RV pacing impedance results were reported at implant
Time Frame: implant
Population: 79 CRT-D and 46 ICD patients had data available at implant
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 79 | 46
Ohms | 637 (208) | 807 (385)

24. Primary Outcome: Clinical Performance at Pre-discharge for RV Pacing Impedance
Description: RV pacing impedance results were reported for pre-discharge
Time Frame: pre-discharge
Population: 78 CRT-D and 45 ICD patients had data available at pre-discharge
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 78 | 45
Ohms | 604 (196) | 686 (284)

25. Primary Outcome: Clinical Performance at 1-month for RV Pacing Impedance
Description: RV pacing impedance results were reported at 1-month post-implant
Time Frame: 1-month
Population: 75 CRT-D and 43 ICD patients had data available at 1-month visit
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 75 | 43
Ohms | 590 (209) | 658 (295)

26. Primary Outcome: Clinical Performance at Implant for RA Pacing Impedance
Description: RA pacing impedance results were reported at implant
Time Frame: implant
Population: 56 CRT-D and 11 ICD patients had data available at implant
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 56 | 11
Ohms | 538 (132) | 670 (443)

27. Primary Outcome: Clinical Performance at Pre-discharge for RA Pacing Impedance
Description: RA pacing impedance results were reported at pre-discharge
Time Frame: pre-discharge
Population: 57 CRT-D and 11 ICD patients had data available at pre-discharge
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 57 | 11
Ohms | 512 (141) | 656 (448)

28. Primary Outcome: Clinical Performance at 1-month for RA Pacing Impedance
Description: RA pacing impedance results were reported at 1-month post-implant
Time Frame: 1-month
Population: 54 CRT-D and 11 ICD patients had data available at 1-month
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | INCEPTA CRT-D Patients | INCEPTA ICD Patients
Number analyzed (Participants) | 54 | 11
Ohms | 534 (152) | 655 (447)

29. Primary Outcome: Product Experiences Reported by the Site for All Patients for Study Duration
Description: Product experiences reported may include the shock impedance noise display, problems encountered with the universal serial bus (USB), a program parameter mismatch, reverse mode switches, electrogram (EGM) noise without oversensing, lead connection issues, or customer device feedback.
Time Frame: Overall study results
Population: All patients from overall study population were considered. Of the total population, the number of product experiences was reported.
Measure: Number; unit: experiences
Arm/Group | INCEPTA CRT-D and ICD Patients (Overall Study Population)
Number analyzed (Participants) | 120
experiences | 65

30. Primary Outcome: Induced Ventricular Tachycardia / Ventricular Fibrillation (VT/VF) Episode Successful Conversion Rates at Implant
Description: The % of successful conversions after inducing a VT/VF episode was analyzed for available data from CRT and ICD group patients. All episodes of induced VT/VF that resolved with successful conversion were counted from the total attempted conversions and reported as the % of successful conversions from those attempted.
Time Frame: implant
Population: Of the 30 CRT-D and 22 ICD patients with induced episodes, the number with successful conversions was determined. The % of patients that had successful conversion was then reported.
Measure: Number; unit: percentage of successful conversions
Arm/Group | INCEPTA CRT-D | INCEPTA ICD
Number analyzed (Participants) | 30 | 22
percentage of successful conversions | 100 | 100

31. Primary Outcome: Induced VT/VF Episode Successful Conversion Rates at 1-month
Description: as for outcome 30
Time Frame: 1-month
Population: Of all patients that experienced an induced VT/VF episode at 1-month, the number that had successful conversions was reported for both CRT-D and ICD patients.
Measure: Number; unit: percentage of successful conversions
Arm/Group | INCEPTA CRT-D | INCEPTA ICD
Number analyzed (Participants) | 1 | 1
percentage of successful conversions | 100 | 100

32. Primary Outcome: Induced VT/VF Episode Successful Conversion Rates at 3-months
Description: as for outcome 30
Time Frame: 3-month
Population: Of the 6 CRTD and 3 ICD patients that had induced VT/VF episodes at 3-month follow-up, the number of those that were converted successfully was reported in %
Measure: Number; unit: percentage of successful conversions
Arm/Group | INCEPTA CRT-D | INCEPTA ICD
Number analyzed (Participants) | 6 | 3
percentage of successful conversions | 100 | 100

33. Primary Outcome: Induced Episode Detection Times at Implant
Description: The mean time it took to complete a successful conversion after inducing a VT/VF episode was analyzed for available data from CRT and ICD group patients. The time was recorded (in seconds) for the time duration that was required to successfully convert the patient after inducing VT/VF.
Time Frame: implant
Population: Of the 30 CRT-D and 22 ICD patients with induced VT/VF episodes, the mean time required for conversion was reported for all available data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | INCEPTA CRT-D | INCEPTA ICD
Number analyzed (Participants) | 30 | 22
seconds | 2.46 (0.38) | 2.40 (0.42)

34. Primary Outcome: Induced Episode Detection Times at 1-month
Description: as for outcome 33
Time Frame: 1-month
Population: Of the 1 CRT-D and 1 ICD patients that underwent induced VT/VF at 1month, the mean time for successful conversion was reported.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | INCEPTA CRT-D | INCEPTA ICD
Number analyzed (Participants) | 1 | 1
seconds | 2.06 (0) | 2.06 (0)

35. Primary Outcome: Induced Episode Detection Times at 3 Months
Description: as for outcome 33
Time Frame: 3-month
Population: Of the 6 CRT-D and 3 ICD patients with available data that had succesful conversion after induced VT/VF episodes, the mean time was determined at 3 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | INCEPTA CRT-D | INCEPTA ICD
Number analyzed (Participants) | 6 | 3
seconds | 2.28 (0.28) | 2.29 (0.06)

36. Primary Outcome: Spontaneous Episode Conversion Success Rate at 3 Months
Description: Of the total patients that experienced a spontaneous episode, the % of patients with a spontaneous rhythm conversion that was successful was determined.
Time Frame: 3-month
Population: Of the 13 CRT-D and 8 ICD patients that experienced a spontaneous episode, the successful conversions were reported.
Measure: Number; unit: percentage of successful conversions
Units Other Than Participants: Number of episodes
Arm/Group | INCEPTA CRT-D | INCEPTA ICD
Number analyzed (Participants) | 13 | 8
Number analyzed (Number of episodes) | 54 | 42
percentage of successful conversions | 100 | 100

37. Primary Outcome: Wanded Telemetry Issues at Pre-discharge Follow-up
Description: The Investigators completed a questionnaire based on the performance of the wanded telemetry during device interrogations at pre-discharge follow-up. The number of problems reported were counted from the entire study cohort.
Time Frame: Pre-Discharge visit occurred after implant but prior to 1 month follow-up visit
Population: 118 was the total number of questionnaires completed and available from the PI for analysis.
Measure: Number; unit: issues
Arm/Group | INCEPTA CRT-D and ICD (Overall Study Population)
Number analyzed (Participants) | 118
issues | 1

ADVERSE EVENTS:
Time Frame: 9 months (with a window of plus/minus 1 month)
Arm/Group | INCEPTA ICD and CRT-D
Serious Adverse Events (participants affected / at risk) | 13/120
Other Adverse Events (participants affected / at risk) | 10/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCEPTA ICD and CRT-D (N=120)
Lead Dislodgement, Left Ventricle (Cardiac disorders) | 2 (3)
Lead Dislodgement, Right Atrium (Cardiac disorders) | 2 (2)
Lead Dislodgement, Right Ventricle (Cardiac disorders) | 2 (2)
Elevated Threshold, Right Atrium (Cardiac disorders) | 1 (1)
Elevated Threshold, Right Ventricle (Cardiac disorders) | 2 (2)
Insulation Breach, Right Atrium (Cardiac disorders) | 1 (1)
Inadvertent Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Unable to Convert, Defibrillation Lead (Cardiac disorders) | 1 (1)
Infection, Post-Surgical (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCEPTA ICD and CRT-D (N=120)
Extra Cardiac Stimulation, Left Ventricle (Cardiac disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall be provided with copy of all Trial-related manuscripts and reports for review and comment